CLINICAL TRIAL: NCT01716533
Title: A Serological Study in Adult Subjects With Clostridium Difficile Infection
Brief Title: Evaluation of the Immune Response to Clostridium Difficile in Adults With Clostridium Difficile Infection (CDI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 116509
Record Dates: First submitted 2012-10-18; First posted 2012-10-30 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-02

CONDITIONS: Infections, Clostridium Difficile
Keywords: Serological; Adults; Clostridium difficile; Adult CDI patients
MeSH Terms: conditions — Clostridium Infections | interventions — Blood Specimen Collection

ARMS (4):
- Recurrence group (Other): Male or female subjects aged 18 years or older at the time of enrollment, who experienced recurrence of Clostridium difficile infection (CDI) after clinical response to antibiotic treatment to treat the initial CDI episode.
  Interventions: Procedure: Blood sampling; Other: Stool sample collection
- Sustained response group (Other): Male or female subjects aged 18 years or older at the time of enrollment, who did not experience recurrence of CDI after clinical response to the antibiotic treatment to treat the initial CDI episode.
  Interventions: Procedure: Blood sampling; Other: Stool sample collection
- Failure to antibiotic Group (Other): Male or female subjects aged 18 years or older at the time of enrollment, withdrawn due to failure of antibiotic treatment to treat the initial CDI episode.
  Interventions: Procedure: Blood sampling; Other: Stool sample collection
- Unclassified Group (Other): Male or female subjects aged 18 years or older at the time of enrollment, who couldn't be classified as sustained response, recurrence, or failure to antibiotic due to missing data.
  Interventions: Procedure: Blood sampling; Other: Stool sample collection

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling will be done at Day 0, at Day 14, at recurrence (if applicable) and at end of follow-up.
Other: Stool sample collection — Stool samples will be collected around Day 0, around Day 14 and at recurrence (if applicable).

SUMMARY:
This study aims to 1) evaluate the C. difficile-specific immune response in CDI patients and 2) explore the difference in immune response between the patients with CDI recurrence and those with a sustained clinical response.

DETAILED DESCRIPTION:
Patients with an initial episode of CDI will be followed up for CDI recurrence or sustained clinical response. The subjects will be allocated into 2 groups at the study end:

* Recurrence Group: Subjects who experience recurrence of CDI after clinical response to antibiotic treatment to treat the initial CDI episode.
* Sustained response Group: Subjects who do not experience recurrence of CDI after clinical response to the antibiotic treatment to treat the initial CDI episode.

This protocol has been amended twice to improve recruitment of subjects in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol or/ and subjects who can receive assistance from his/ her legally acceptable representative (LAR) or a designate who can and will comply with the requirements of the protocol.
* A male or female aged 18 years or older at the time of enrolment.
* Written informed consent obtained from the subject/ LAR of the subject.
* A reasonable prognosis of survival during the study period as judged by the investigator.
* Outpatients, emergency room and/ or hospitalized subjects diagnosed with CDI for which the symptoms started maximum 14 days prior to study enrolment.
* Subjects who receive or plan to receive antibiotic treatment to treat the CDI episode.

Exclusion Criteria:

* Concurrently participating or planning to participate in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous CDI episode within the previous 6 months before study enrolment (except for up to ~25% of the subjects).
* Chronic diarrheal illness such as, but not limited to, ulcerative colitis or Crohn's disease.
* Planned surgery for CDI within 24 hours after study entry.
* Previous vaccination against Clostridium difficile.
* Having received a Clostridium difficile monoclonal antibody product(s) within the previous 3 months or planned administration during the study period.
* Administration of immunoglobulins within the previous 3 months or planned administration during the study period.
* Subject having any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the subject participating in the study, would make it unlikely for the subject to complete the study, or would confound the results of the study.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within the previous 6 months.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history.
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-02-02 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (3):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Houston, Texas
- Canada (2):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 57 subjects were enrolled, among which 11 subjects from one centre in the United States (University of Texas School of Public Health, Houston) who were excluded from final analysis due to GCP issues.
Pre-assignment Details: Two extra groups were identified in addition to the two groups foreseen in the protocol: Failure to antibiotic Group and Unclassified Group.
Groups:
- Recurrence Group: Male or female subjects aged 18 years or older at the time of enrolment, who experienced recurrence of Clostridium difficile infection (CDI) after clinical response to antibiotic treatment to treat the initial CDI episode.
- Sustained Response Group: Male or female subjects aged 18 years or older at the time of enrolment, who did not experience recurrence of CDI after clinical response to the antibiotic treatment to treat the initial CDI episode.
- Failure to Antibiotic Group: Male or female subjects aged 18 years or older at the time of enrolment, withdrawn due to failure of antibiotic treatment to treat the initial CDI episode.
- Unclassified Group: Male or female subjects aged 18 years or older at the time of enrolment, who couldn't be classified as sustained response, recurrence, or failure to antibiotic due to missing data.
Period: Overall Study
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Started | 7 | 25 | 5 | 9
Completed | 7 | 25 | 0 | 1
Not Completed | 0 | 0 | 5 | 8
Not completed — Failure of antibiotic treatment to treat | 0 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 0 | 2
Not completed — Immunosuppressants>14days past 6months | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group | Total
Number analyzed (Participants) | 7 | 25 | 5 | 9 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (18.3) | 53.5 (20.1) | 58.0 (12.0) | 64.0 (18.0) | 55.1 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 16 | 2 | 4 | 25
  Male | 4 | 9 | 3 | 5 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 0 | 4 | 3 | 4 | 11
  Asian - Japanese Heritage | 0 | 1 | 0 | 0 | 1
  Asian - South East Asian Heritage | 0 | 0 | 0 | 1 | 1
  White - Caucasian / European Heritage | 7 | 18 | 2 | 4 | 31
  Unspecified | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Serum Anti-toxin A and Anti-toxin B Antibody Concentrations at Day 14
Description: Serum anti-toxin B antibody concentrations were expressed as Geometric Mean Concentrations (GMCs), as measured by the Enzyme Linked Immunosorbent Assay (ELISA) for the cut-off of equal to or above (≥) 100 EU/mL.
Time Frame: At Day 14
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom the result of the considered assay was available for the blood sample taken at Day 14. The development of the serum anti-toxin A ELISA was cancelled, therefore this analysis was not performed.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 21 | 0 | 2
EU/mL | 2083.3 [995.8 to 4358.5] | 3189.4 [1338.4 to 7600.2] |  | 32096.4 [26.1 to 39518495]
Statistical Analysis 1: Comparison: Recurrence Group vs Sustained Response Group; ELISA anti-toxin B antibody concentrations at Day 14 were compared between the Sustained response Group and Recurrence Group by using a one-way analysis of variance (ANOVA) model on the log-transformed concentration; Test type: Superiority; p = 0.5746, ANOVA — P-value = two-sided p-value for HO: GMC ratio = 1 (ANOVA model, T-test), groups considered as statistically significant different if the two-sided p-value is below 0.05; ANOVA model -pooled variance; GMC ratio = 1.53, 95% CI 2-sided [0.33 to 7.14] — GMC ratio = GMC Sustained response Group /GMC Recurrence Group

2. Primary Outcome: Serum F2 C-terminal Anti-toxin B Antibody Concentrations
Description: Serum F2 C-terminal anti-toxin B antibody concentrations were expressed as Geometric Mean Concentrations (GMCs), as measured by ELISA for the cut-off of 13.16 EU/mL.
Time Frame: At Day 14
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom the result of the considered assay was available for the blood sample taken at Day 14.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 20 | 0 | 2
EU/mL | 149.3 [20.2 to 1102.9] | 246.6 [52.7 to 1154.8] |  | 10736.7 [1.7 to 69276208]
Statistical Analysis 1: Comparison: Recurrence Group vs Sustained Response Group; Serum F2 C-terminal anti-toxin B antibody concentrations at Day 14 were compared between the Sustained response Group and Recurrence Group by using a one-way analysis of variance (ANOVA) model on the log-transformed concentration; Test type: Superiority — ANOVA model -pooled variance; p = 0.7124, ANOVA — P-value = two-sided p-value for HO: GMC ratio = 1, groups considered as statistically significant different if the two-sided p-value is below 0.05; GMC ratio = 1.65, 95% CI 2-sided [0.10 to 26.41] — GMC ratio = GMC Sustained response Group /GMC Recurrence Group

3. Secondary Outcome: Serum Anti-toxin A and Anti-toxin B Antibody Concentrations at Day 0 and Day 72
Description: Serum anti-toxin B antibody concentrations were expressed as Geometric Mean Concentrations (GMCs), as measured by ELISA for the cut-off equal to or above (≥) 100 EU/mL.
Time Frame: At Day 0 and at Day 72
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom the result of at least one assay was available for the blood sample taken at Day 72. The development of the serum anti-toxin A ELISA was cancelled, therefore this analysis was not performed.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 22 | 0 | 2
EU/mL
  Anti-toxin B at Day 0 | 1939.6 [847.2 to 4440.6] | 1682.9 [858.7 to 3298.2] |  | 19638.5 [217.5 to 1773406]
  Anti-toxin B at Day 72: number analyzed (Participants) | 7 | 22 | 0 | 1
  Anti-toxin B at Day 72 | 4471.1 [1441.1 to 13871.8] | 3670.4 [1519.8 to 8864.6] |  | 64050.6 [NA to NA] — Upper and lower limits were not available as there was only one subject assessed for this time point.

4. Secondary Outcome: Serum Neutralizing Anti-toxin A and Anti-toxin B Antibody Titers at Day 14
Description: Neutralizing antibody concentrations were expressed as Geometric Mean Titers (GMTs), as measured in an inhibition of cytotoxicity assay (toxin neutralization assays) for the cut-off of 2, expressed in 1/DIL unit, in which DIL is the sample dilution corresponding to 50% neutralization.
Time Frame: At Day 14
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom the result of at least one assay was available for the blood sample taken at Day 14.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 22 | 0 | 2
Titer
  Neutralizing anti-toxin A: number analyzed (Participants) | 7 | 19 | 0 | 2
  Neutralizing anti-toxin A | 11.3 [0.7 to 194.8] | 2.3 [1.2 to 4.5] |  | 4.7 [0.0 to 1584000000]
  Neutralizing anti-toxin B | 2.7 [0.4 to 18.2] | 15.3 [4.2 to 55.1] |  | 1725.7 [125.5 to 23728.0]

5. Secondary Outcome: Serum Neutralizing Anti-toxin A and Anti-toxin B Antibody Titers at Day 0, Within 10 Days After Recurrence and at Day 72
Description: Neutralizing antibody concentrations were expressed as Geometric Mean Titers (GMTs), as measured in an inhibition of cytotoxicity assay (toxin neutralization assays) for the cut-off of 2, expressed in 1/DIL unit, in which DIL is the sample dilution corresponding to 50% neutralization. This measure concerned only diarrhea recurrence. No CDI recurrence was considered as part of the Group Sustained Response.
Time Frame: At Day 0, within 10 days after start of recurrent episode if any, and at end of follow-up (Day 72)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom the result for the considered assay was available for the blood sample taken at the considered time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 25 | 0 | 7
Titer
  Neutralizing anti-toxin A, Day 0: number analyzed (Participants) | 6 | 19 | 0 | 2
  Neutralizing anti-toxin A, Day 0 | 14.8 [0.4 to 525.0] | 1.5 [0.9 to 2.4] |  | 3.2 [0.0 to 7130211]
  Neutralizing anti-toxin A, recurrence 1: number analyzed (Participants) | 7 | 1 | 0 | 0
  Neutralizing anti-toxin A, recurrence 1 | 12.2 [0.6 to 241.2] | 1.0 [NA to NA] — Upper and lower limits were not available as there was only one subject assessed for this time point. |  |
  Neutralizing anti-toxin A, recurrence 2: number analyzed (Participants) | 1 | 0 | 0 | 0
  Neutralizing anti-toxin A, recurrence 2 | 1.0 [NA to NA] — Upper and lower limits were not available as there was only one subject assessed for this time point. |  |  |
  Neutralizing anti-toxin A, Day 72: number analyzed (Participants) | 6 | 20 | 0 | 0
  Neutralizing anti-toxin A, Day 72 | 11.1 [0.3 to 422.0] | 2.5 [1.2 to 5.4] |  |
  Neutralizing anti-toxin B, Day 0: number analyzed (Participants) | 6 | 21 | 0 | 2
  Neutralizing anti-toxin B, Day 0 | 3.3 [0.4 to 28.0] | 9.6 [2.7 to 34.1] |  | 340.3 [0.0 to 461890000]
  Neutralizing anti-toxin B, recurrence 1: number analyzed (Participants) | 7 | 1 | 0 | 0
  Neutralizing anti-toxin B, recurrence 1 | 3.0 [0.4 to 22.3] | 1.0 [NA to NA] — Upper and lower limits were not available as there was only one subject assessed for this time point. |  |
  Neutralizing anti-toxin B, recurrence 2: number analyzed (Participants) | 1 | 0 | 0 | 0
  Neutralizing anti-toxin B, recurrence 2 | 1.0 [NA to NA] — Upper and lower limits were not available as there was only one subject assessed for this time point. |  |  |
  Neutralizing anti-toxin B, Day 72: number analyzed (Participants) | 7 | 22 | 0 | 1
  Neutralizing anti-toxin B, Day 72 | 8.0 [1.1 to 56.8] | 16.2 [4.3 to 60.3] |  | 1372.0 [NA to NA] — Upper and lower limits were not available as there was only one subject assessed for this time point.

6. Secondary Outcome: Number of Subjects With Clostridium Difficile Infection (CDI) Recurrence
Description: A CDI recurrence is defined as the development of a new episode of CDI following clinical response at the end of standard of care (SoC) for the initial CDI episode.
Time Frame: From Day 0 to Day 72
Population: The analysis was performed on the Total enrolled cohort, which included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 25 | 5 | 9
Participants | 7 | 0 | 0 | 0

7. Secondary Outcome: CDI Initial Episodes Severity Characteristics, in All Subjects
Description: Severity characteristics were expressed in duration of days for hospitalization, intensive care unit, Standard of Care (SoC) and CDI episodes.
Time Frame: At Day 0
Population: The analysis was performed on the Total enrolled cohort, which included all subjects enrolled in the study and who reported any of the characteristics assessed.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 25 | 5 | 9
Days
  Duration of hospitalization: number analyzed (Participants) | 0 | 10 | 1 | 7
  Duration of hospitalization |  | 5.0 [4.0 to 11.0] | 7.0 [7.0 to 7.0] | 16.0 [8.0 to 22.0]
  Duration in intensive care unit: number analyzed (Participants) | 0 | 2 | 0 | 3
  Duration in intensive care unit |  | 5.0 [4.0 to 6.0] |  | 8.0 [7.0 to 17.0]
  Duration of CDI episodes: number analyzed (Participants) | 4 | 13 | 4 | 2
  Duration of CDI episodes | 10.5 [9.0 to 15.0] | 6.0 [4.0 to 13.0] | 24.0 [14.5 to 33.5] | 10.0 [5.0 to 15.0]
  Duration of SoC: number analyzed (Participants) | 7 | 25 | 3 | 3
  Duration of SoC | 11.0 [11.0 to 15.0] | 14.0 [11.0 to 16.0] | 34.0 [11.0 to 84.0] | 11.0 [10.0 to 26.0]

8. Secondary Outcome: Number of Subjects With Initial CDI Episode by Severity, in All Subjects
Description: Initial CDI episodes were recorded by severity criteria: medical attention given, admission to intensive care unit, colectomy, death, high white blood cells (WBC) count, high creatinine count, hypotension/shock, clinical response to Standard of Care (SoC).
Time Frame: At Day 0
Population: The analysis was performed on the Total enrolled cohort, which included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 25 | 5 | 9
Participants
  Medical attention - Medical contact without visit | 1 | 1 | 1 | 0
  Medical attention - Medical personnel visit | 2 | 3 | 1 | 0
  Medical attention - Emergency Room | 2 | 6 | 1 | 1
  Medical attention - Hospitalization | 2 | 15 | 2 | 8
  Intensive care unit - Yes | 0 | 3 | 0 | 3
  Intensive care unit - No | 7 | 22 | 5 | 6
  Colectomy - Yes | 0 | 0 | 0 | 0
  Colectomy - No | 7 | 25 | 5 | 9
  Death - Yes | 0 | 0 | 0 | 0
  Death - No | 7 | 25 | 5 | 9
  Non-severe CDI episode | 7 | 23 | 5 | 6
  Severe CDI episode | 0 | 2 | 0 | 3
  Leukocytosis with high WBC count: number analyzed (Participants) | 0 | 2 | 0 | 3
  Leukocytosis with high WBC count | 0 | 1 | 0 | 1
  Serum creatinine high level: number analyzed (Participants) | 0 | 2 | 0 | 3
  Serum creatinine high level | 0 | 0 | 0 | 1
  Hypotension/shock: number analyzed (Participants) | 0 | 2 | 0 | 3
  Hypotension/shock | 0 | 0 | 0 | 1
  Leukocytosis with high WBC count+Hypotension/shock: number analyzed (Participants) | 0 | 2 | 0 | 3
  Leukocytosis with high WBC count+Hypotension/shock | 0 | 1 | 0 | 0
  Clinical response at end of SoC - Yes | 6 | 18 | 0 | 1
  Clinical response at end of SoC - No | 1 | 4 | 2 | 1
  Clinical response at end of SoC - Unspecified | 0 | 3 | 3 | 7
  Detection of C. difficile strains - Yes | 1 | 2 | 0 | 1
  Detection of C. difficile strains - No | 6 | 23 | 5 | 5
  Stool not collected or discarded - CDI detection | 0 | 0 | 0 | 3

9. Secondary Outcome: Number of Subjects With CDI Recurrence by Severity, in Those Subjects Who Recur
Description: A CDI recurrence is defined as the development of a new episode of CDI following clinical response at the end of standard of care (SoC) for the initial CDI episode. An episode of diarrhea was not considered as a recurrence of CDI if the stool was negative for C. difficile or if the diarrhea was attributed to another cause than C. difficile. The severity criteria for CDI recurrent episodes were categorized into non-severe and severe.
Time Frame: At recurrence (within 10 days of start diarrhea) during a follow up period of up to 72 days per participant
Population: The analysis was performed on the Total enrolled cohort, which included all subjects enrolled in the study who recurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 0 | 0 | 0
Participants
  Non-severe | 7 |  |  |
  Severe | 0 |  |  |

10. Secondary Outcome: Number of Subjects With Failure of Antibiotic Treatment
Description: Failure of antibiotic treatment against C. difficile is defined as the persistence or the incomplete resolution of symptoms (more than one unformed stool per day) after a full course of antibiotic(s) therapy (minimum 7 days).
  Aminopen+BetaLactam Inhib,1st Gen.Cephalosporin = Aminopenicillin+Beta-Lactamase Inhibitor and 1st Generation Cephalosporin.
  Aminopen+BetaLactam Inhib, 3rd Gen.Cephalosporin = Aminopenicillin+Beta-Lactamase Inhibitor and 3rd Generation Cephalosporin excluding Ceftazidime and Fluoroquinolone.
  Aminopen+BetaLactam Inhib and Fluoroquinolone = Aminopenicillin+Beta-Lactamase Inhibitor and Fluoroquinolone.
  Antipseudom Pen+BetaLactam Inhib and Cephalosporin = Antipseudomonal Penicillin+Beta-Lactamase Inhibitor and 1st Generation Cephalosporin and 3rd Generation Cephalosporin excluding Ceftazidime and Fluoroquinolone and Glycopeptides (Iv).
  Antipseudom Pen+BetaLactam Inhib and Glycopeptides = Antipseudomonal Penicillin+Beta-Lactamase Inhibitor and Glycopeptides (Iv).
Time Frame: Within 3 months before the initial CDI episodes
Population: The analysis was performed on the Total enrolled cohort, which included all evaluable subjects for whom results about failure of antibiotic treatment (not prescribed to treat Clostridium difficile) were available within 3 months before the initial CDI episodes.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 6 | 18 | 2 | 6
Participants
  1st Generation Cephalosporin | 0 | 2 | 1 | 0
  1st Gen Cephalosporin+Tetracyclin, no Tigecyclin | 1 | 0 | 0 | 0
  3rd Generation Cephalosporin, no Ceftazidime | 0 | 1 | 0 | 0
  4th Generation Cephalosporin and Fluoroquinolone | 0 | 1 | 0 | 0
  Aminopenicillin | 0 | 3 | 0 | 0
  Aminopen+BetaLactam Inhib,1st Gen.Cephalosporin | 1 | 0 | 0 | 0
  Aminopen+BetaLactam Inhib, 3rd Gen.Cephalosporin | 1 | 0 | 0 | 0
  Aminopen+BetaLactam Inhib and Fluoroquinolone | 0 | 0 | 0 | 1
  Aminopenicillin And Macrolide | 0 | 1 | 0 | 0
  Antipseudom Pen+BetaLactam Inhib and Cephalosporin | 0 | 0 | 0 | 1
  Antipseudom Pen+BetaLactam Inhib and Glycopeptides | 0 | 0 | 0 | 1
  Fluoroquinolone | 0 | 1 | 1 | 1
  Fluoroquinolone And 3rd/4th Gen Fluoroquinolone | 0 | 1 | 0 | 0
  Fluoroquinolone And Lincosamide | 0 | 1 | 0 | 0
  Glycopeptides (Iv) | 0 | 1 | 0 | 1
  Lincosamide | 2 | 1 | 0 | 0
  Macrolide | 0 | 1 | 0 | 0
  Metronidazole and Aminopenicillin | 0 | 1 | 0 | 0
  Metronidazole and Fluoroquinolone and Lincosamide | 1 | 0 | 0 | 0
  Monobactam And Fluoroquinolone | 0 | 1 | 0 | 0
  Rifamycin | 0 | 1 | 0 | 1
  Subject Does Not Recall Name Of Abx | 0 | 1 | 0 | 0

11. Secondary Outcome: Number of Subjects With Risk Factors Associated With the Initial CDI Episode
Description: Risk factors for CDI included factors in three main domains involving host factors (advanced age, impaired immune status, co-morbidities); increased exposure to C. difficile spores (longer length of stays, healthcare environment, infected roommates or hand carriage by personnel); and factors that disrupt the normally protective colonic microflora layer (antimicrobials, other medications or procedures).
  CDI episodes within 6 months: Protocol exclusion criteria for enrolment allowed up to maximum 25% of the planned subjects having a previous CDI episode within the previous 6 months.
  Antibiotic taken within 3 months: Antibiotic not prescribed to treat C. difficile taken within 3 months before the current CDI episode.
Time Frame: At Day 0
Population: The analysis was performed on the Total enrolled cohort, which included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 25 | 5 | 9
Participants
  Setting of CDI development: Community | 5 | 18 | 3 | 2
  Setting of CDI development: Hospital | 2 | 6 | 1 | 6
  Setting of CDI development: Nursing home | 0 | 0 | 0 | 0
  Setting of CDI development: Rehabilitation center | 0 | 0 | 0 | 0
  Setting of CDI development: Other | 0 | 1 | 1 | 1
  No CDI episodes within 6 months | 6 | 22 | 4 | 8
  CDI episodes within 6 months | 1 | 3 | 1 | 1
  No admission to hospital within 3 months | 6 | 15 | 4 | 4
  Admission to hospital within 3 months | 1 | 10 | 1 | 5
  Not staying in nursing home within 3 months | 7 | 25 | 5 | 8
  Staying in nursing home within 3 months | 0 | 0 | 0 | 1
  Not staying in rehabilitation center within 3 mths | 7 | 25 | 5 | 8
  Staying in rehabilitation center within 3 months | 0 | 0 | 0 | 1
  No antibiotic taken within 3 months | 1 | 7 | 3 | 3
  Antibiotic taken within 3 months | 6 | 18 | 2 | 6
  No proton Pump Inhibitors taken within 3 months | 2 | 18 | 0 | 4
  Proton Pump Inhibitors taken within 3 months | 5 | 7 | 5 | 5
  No anti-acid drugs taken within 3 months | 3 | 24 | 4 | 7
  Anti-acid drugs taken within 3 months | 4 | 1 | 1 | 2
  No nutrition via feeding tube within 3 months | 7 | 25 | 5 | 9
  Nutrition via feeding tube within 3 months | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Subjects With Risk Factors Associated With the CDI Recurrence
Description: Risk factors for CDI included factors in three main domains involving host factors (advanced age, impaired immune status, co-morbidities); increased exposure to C. difficile spores (longer length of stays, healthcare environment, infected roommates or hand carriage by personnel); and factors that disrupt the normally protective colonic microflora layer (antimicrobials, other medications or procedures).
Time Frame: At recurrence (within 10 days of start diarrhea) during a follow up period of up to 72 days per participant
Population: The analysis was performed on the Total enrolled cohort, which included all subjects enrolled in the study who recurred.
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
Number analyzed (Participants) | 7 | 0 | 0 | 0
Participants
  Setting of CDI development: Community | 6 |  |  |
  Setting of CDI development: Hospital | 1 |  |  |
  Setting of CDI development: Nursing home | 0 |  |  |
  Setting of CDI development: Rehabilitation center | 0 | 0 |  |
  Setting of CDI development: Other | 0 |  |  |
  No admission to hospital during follow-up period | 7 |  |  |
  Admission to hospital during follow-up period | 0 |  |  |
  Not staying in nursing home during FU period | 7 |  |  |
  Staying in nursing home during follow-up period | 0 |  |  |
  Not staying in rehab. center during FU period | 7 |  |  |
  Staying in rehabilitation center during FU period | 0 |  |  |
  No antibiotic taken during FU period | 5 |  |  |
  Antibiotic taken during FU period | 2 |  |  |
  No Proton Pump Inhibitors taken during FU period | 4 |  |  |
  Proton Pump Inhibitors taken during FU period | 3 |  |  |
  No anti-acid drugs taken during FU period | 6 |  |  |
  Anti-acid drugs taken during FU period | 1 |  |  |
  No nutrition via feeding tube during FU period | 7 |  |  |
  Nutrition via feeding tube during FU period | 0 |  |  |

ADVERSE EVENTS:
Time Frame: Serious adverse events related to study participation or to a concurrent GSK medication/vaccine were collected during the entire study period (from Day 0 to Day 72).
Description: Only SAEs related to study participation or to a concurrent GSK medication/vaccine were collected as part of this study. The fatal events observed were not considered to be related to study participation nor to a concurrent GSK medication/vaccine, and are reported in the Participant Flow section in addition to the All-Cause Mortality Section. No other adverse events were collected during the study period.
Arm/Group | Recurrence Group | Sustained Response Group | Failure to Antibiotic Group | Unclassified Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/25 | 0/5 | 2/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/25 | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.